CLINICAL TRIAL: NCT04735432
Title: A Phase 3, Randomized, Open-Label, Parallel-Group Study to Compare the Pharmacodynamics, Pharmacokinetics, Efficacy, Safety, Tolerability, and Immunogenicity of Multiple Subcutaneous Injections of Efgartigimod PH20 SC With Multiple Intravenous Infusions of Efgartigimod in Patients With Generalized Myasthenia Gravis
Brief Title: Evaluating the Pharmacodynamic Noninferiority of Efgartigimod PH20 SC Administered Subcutaneously as Compared to Efgartigimod Administered Intravenously in Patients With Generalized Myasthenia Gravis
Acronym: ADAPTsc
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2001
Record Dates: First submitted 2021-01-26; First posted 2021-02-03 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-01

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- efgartigimod PH20 SC (Experimental): Patients receiving efgartigimod PH20 subcutaneous (SC) treatment
  Interventions: Biological: efgartigimod PH20 SC
- efgartigimod (Experimental): Patients receiving efgartigimod intravenous (IV) treatment
  Interventions: Biological: efgartigimod IV

INTERVENTIONS:
Biological: efgartigimod PH20 SC — Subcutaneous injection with efgartigimod PH20 SC
  Arms: efgartigimod PH20 SC
Biological: efgartigimod IV — Intravenous infusion of efgartigimod
  Arms: efgartigimod

SUMMARY:
The purpose of this study is to investigate the Pharmacodynamics (PD), Pharmacokinetics (PK), safety, tolerability, immunogenicity, and clinical efficacy of efgartigimod coformulated with recombinant human hyaluronidase PH20 (rHuPH20) as compared to efgartigimod IV infused in patients with generalized myasthenia gravis (gMG). The study duration is approximately 12 weeks. After screening, patients will be randomized to receive either efgartigimod infusions or efgartigimod PH20 subcutaneously (SC)

DETAILED DESCRIPTION:
Main objective of the trial: To demonstrate that the pharmacodynamic (PD) effect of injections of 1000 mg efgartigimod PH20 SC (efgartigimod co-formulated with recombinant humanhyaluronidase PH20 for subcutaneous administration), administered once weekly for 4 administrations, is NI (noninferior) to IV infusions of efgartigimod (efgartigimod formulation for intravenous infusion) at a dose of 10 mg/kg administered once weekly for 4 administrations.

Secondary objectives: To compare the PD effect of efgartigimod PH20 SC and efgartigimod IV over time; To evaluate the pharmacokinetics (PK) of efgartigimod PH20 SC and efgartigimod IV; To evaluate the safety, tolerability, and immunogenicity of efgartigimod PH20 SC and efgartigimod IV; To evaluate the clinical efficacy of efgartigimod PH20 SC and efgartigimod IV.

ELIGIBILITY:
Inclusion Criteria:

Bullet list of each inclusion criterium:

1. Must be capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. At least 18 years of age at the time of signing the informed consent form.
3. Diagnosed with generalized Myasthenia Gravis (gMG) with confirmed documentation and supported by at least 1 of the following:

   1. History of abnormal neuromuscular transmission demonstrated by single fiber electromyography or repetitive nerve stimulation
   2. History of positive edrophonium chloride test
   3. Demonstrated improvement in Myasthenia Gravis (MG) signs upon treatment with oral acetylcholinesterase (AChE) inhibitors as assessed by the treating physician
4. Meeting the clinical criteria as defined by the Myasthenia Gravis Foundation of America (MGFA) class II, III, IVa, or IVb

Exclusion Criteria:

Bullet list of each exclusion criterium:

1. Are pregnant or lactating, or intend to become pregnant during the study or within 90 days after the last dose of Investigational Medicinal Product.
2. Has any of the following medical conditions:

   1. Clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection at screening
   2. Any other known autoimmune disease that, in the opinion of the investigator, would interfere with an accurate assessment of clinical symptoms of myasthenia gravis or put the participant at undue risk.
   3. History of malignancy unless deemed cured by adequate treatment with no evidence of reoccurrence for ≥3 years before the first administration of the IMP. Participants with the following cancers can be included at any time:

      * adequately treated basal cell or squamous cell skin cancer
      * carcinoma in situ of the cervix
      * carcinoma in situ of the breast
      * incidental histological findings of prostate cancer (TNM Classification of Malignant Tumors stage T1a or T1b).
   4. Clinical evidence of other significant serious diseases, or the participant has had a recent major surgery, or who have any other condition that, in the opinion of the investigator, could confound the results of the study or put the participant at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (14):
  - Investigator site 2 - US0010032, Carlsbad, California
  - Investigator Site 41 - US0010004, Orange, California
  - Investigator site 2 - US0010108, Boca Raton, Florida
  - Investigator site 1 - US0010110, Port Charlotte, Florida
  - Investigator Site 27 - US0010006, Tampa, Florida
  - Investigator Site 47 - US0010113, Augusta, Georgia
  - Investigator Site 42 - US0010015, Kansas City, Kansas
  - Investigator Site 11 - US0010111, Amherst, New York
  - Investigator Site 40 - US0010003, Chapel Hill, North Carolina
  - Investigator Site 38 - US0010077, Durham, North Carolina
  - Investigator Site 43 - 0010019, Cleveland, Ohio
  - Investigator site 4 - US0010008, Cordova, Tennessee
  - Investigator Site 28 - US0010066, Austin, Texas
  - Investigator Site 46 - US0010009, Texas City, Texas
- Investigator site 5 - BE0320007, Ghent, East-Flanders, Belgium
- Georgia (5):
  - Investigator site 13 - GE9950002, Tbilisi
  - Investigator site 12 - GE9950001, Tbilisi
  - Investigator site 14 - GE9950003, Tbilisi
  - Investigator Site 44 - GE9950004, Tbilisi
  - Investigator Site 45 - GE9950016, Tbilisi
- Germany (2):
  - Investigator Site 30 - DE490006, Berlin
  - Investigator Site 29 - DE490009, Münster
- Hungary (2):
  - Investigator site 15 - HU0360013, Budapest
  - Investigator Site 16 - HU0360020, Debrecen
- Italy (2):
  - Investigator Site 17 - IT0390003, Milan
  - Investigator Site 39 - IT0390008, Roma
- Japan (8):
  - Investigator Site 31 - JP0810055, Sapporo, Hokkaido
  - Investigator Site 18 - JP0810002, Chiba
  - Investigator site 6 - JPN0810004, Hanamaki
  - Investigator Site 33 - JP0810058, Hiroshima
  - Investigator Site 19 - JP0810007, Osaka
  - Investigator Site 34 - JP0810005, Sendai
  - Investigator Site 32 - JP0810059, Tokyo
  - Investigator Site 20 - JP0810009, Tokyo
- Investigator Site 7 - NL0310001, Leiden, Netherlands
- Poland (6):
  - Investigator Site 21 - PL0480001, Gdansk
  - Investigator Site 8 - PL0480007, Katowice
  - Investigator Site 9 - PL0480024, Krakow
  - Investigator Site 22 - PL0480005, Krakow
  - Investigator Site 23 - PL0480018, Lublin
  - Investigator Site 24 - PL0480022, Warsaw
- Russia (2):
  - Investigator Site 35 - RU0070002, Novosibirsk
  - Investigator Site 36 - RU0070014, Saint Petersburg
- Spain (4):
  - Investigator Site 37 - ES0340021, Barcelona
  - Investigator Site 26 - ES0340038, Barcelona
  - Investigator Site 25 - ES0340002, Madrid
  - Investigator Site 10 - ES0340039, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant's evaluation of eligibility was performed at screening and confirmed at randomization visit 1. The overall study duration per subject was approximately 12 weeks spanning the study periods - 2 weeks for screening, 3 weeks for treatment, and 7 weeks for follow-up.
Pre-assignment Details: 153 patients were screened, 111 patients were randomized 1:1 to receive efgartigimod PH20 SC 1000 mg (55) or efgartigimod IV 10 mg/kg (56) once weekly for 4 administrations (4 doses on days 1, 8, 15, and 22). 110 patients started in the study (received treatment) as one participant randomized to the efgartigimod IV arm did not receive treatment due to an AE. 55 patients received study treatment in each treatment arm.
Groups:
- Efgartigimod PH20 SC: Patients receiving efgartigimod PH20 subcutaneous (SC) treatment.
  efgartigimod PH20 SC: Subcutaneous injection with 1000 mg efgartigimod PH20 SC
- Efgartigimod IV: Patients receiving 10 mg/kg efgartigimod intravenous (IV) treatment.
  efgartigimod IV: Intravenous infusion of efgartigimod
Period: Overall Study
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Started | 55 | 55
Completed | 52 | 55
Not Completed | 3 | 0
Not completed — Other - due to personal reason | 1 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: ITT analysis set: All randomized participants who were exposed to the IMP. mITT analysis set: All randomized participants with a value for total IgG levels at baseline and at least 1 postbaseline time point. Safety analysis set: All randomized participants who were exposed to IMP. PK analysis set: A subset of the safety analysis set with at least 1 post dose PK measurement.
Groups:
- Efgartigimod PH20 SC: Patients receiving 1000 mg efgartigimod PH20 subcutaneous (SC) treatment.
  efgartigimod PH20 SC: Subcutaneous injection with efgartigimod PH20 SC
- Total: Total of all reporting groups
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 37 | 80
  >=65 years | 12 | 18 | 30
Age, Continuous [Median (Full Range); unit: years] | 53.0 [19 to 84] | 59.0 [24 to 83] | 53.5 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 24 | 21 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 51 | 101
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total IgG Levels at Day 29 (mITT Analysis Set)
Description: ANCOVA Analysis of Percent Change From Baseline in Total IgG Level at Day 29 (ie, 7 days after the fourth IV or SC administration).
Time Frame: From week 0 to week 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 50 | 52
percent | -66.4 [-68.91 to -63.86] | -62.2 [-64.67 to -59.72]
Statistical Analysis 1: Comparison: Efgartigimod PH20 SC vs Efgartigimod IV; The primary endpoint was analyzed using an ANCOVA model with treatment as a factor and total IgG levels at baseline as a covariate. The NI evaluation was based on a percent reduction from baseline in total IgG levels at day 29 (week 4) using an NI margin of 10%. Only the results for mITT analysis set are entered; Test type: Non-Inferiority — This was a phase 3, multicenter, randomized, open-label, parallel-group, 12-week study to evaluate the noninferiority of the pharmacodynamic effect of efgartigimod PH20 SC 1000 mg compared with efgartigimod IV 10 mg/kg in patients with generalized myasthenia gravis; p < 0.0001, ANCOVA; LS mean difference = -4.2, 95% CI 2-sided [-7.73 to -0.66], Standard Error of Mean 1.782

2. Secondary Outcome: Percent Change From Baseline in Total IgG Levels Over Time (mITT Analysis Set)
Description: Total IgG level percent change from baseline over time for the overall population.
Time Frame: From baseline to week 10
Population: mITT Analysis Set: All randomized participants with a value for total IgG levels at baseline and at least 1 postbaseline timepoint.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 55 | 55
percent
  Week 1 | -40.1 (1.45) | -39.6 (1.51)
  Week 2 | -56.9 (1.57) | -55.1 (1.85)
  Week 3 | -62.2 (1.41) | -59 (2)
  Week 4 | -64.7 (1.95) | -62.3 (1.24)
  Week 5 | -57.4 (1.7) | -49.9 (2.17)
  Week 6 | -44 (2.52) | -38.9 (2.24)
  Week 7 | -31.2 (4.67) | -25.3 (2.78)
  Week 8 | -8.9 (8.65) | -14.6 (3.13)
  Week 10 | 7.8 (7.78) | -3.1 (3.82)

3. Secondary Outcome: Percent Change From Baseline in AChR-Ab Levels Over Time in AChR- Ab Positive Patients (mITT Analysis Set)
Description: Percent reduction from baseline in AChR-Ab levels over time in AChR-Ab positive patients measured in mITT Analysis Set.
  Descriptive statistics have been used for this secondary end point.
Time Frame: From baseline to week 10
Measure: Mean (Standard Error); unit: percent
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 45 | 46
percent
  Week 1 | -42.5 (1.5) | -43.7 (1.55)
  Week 2 | -57.4 (1.39) | -55.1 (1.52)
  Week 3 | -61.8 (1.6) | -59.2 (1.66)
  Week 4 | -62.2 (1.76) | -59.6 (1.74)
  Week 5 | -55.3 (1.52) | -47.2 (2.98)
  Week 6 | -40.4 (3.13) | -29.9 (4.61)
  Week 7 | -26.7 (4.76) | -15.8 (5.63)
  Week 8 | -14.5 (7.82) | -7.1 (6.02)
  Week 10 | 13.5 (23.16) | 10.3 (7.85)

4. Secondary Outcome: Percent Change From Baseline in IgG Subtype Levels Over Time (mITT Analysis Set)
Description: Median (IQR) Percent Change From Baseline for the IgG Subtypes (IgG1, IgG2, IgG3, and IgG4) in the Overall Population.
  The highest number of patients among all weeks for the analysis is chosen for each arm.
  Descriptive statistics have been used for this secondary end point.
Time Frame: Baseline to week 10
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 55 | 55
Percent change
  Percent change from baseline at week 4 IgG1 | -71 [-79.3 to -56.6] | -68.4 [-73 to -61.5]
  Percent change from baseline at week 4 IgG2 | -65.6 [-72.2 to -58.1] | -64.5 [-73 to -57.4]
  Percent change from baseline at week 4 IgG3 | -69.6 [-78.3 to -58.4] | -64.7 [-76.9 to -59.5]
  Percent change from baseline at week 4 IgG4 | -56.4 [-64.4 to -37.2] | -55.5 [-64.2 to -42.1]

5. Secondary Outcome: AUEC of the Percent Change From Baseline in Total IgG Level (mITT Analysis Set)
Description: AUEC of the percent reduction from baseline total IgG per dosing interval (days 1-8, days 8-15, days 15-22, and days 22-29), days 1-29, days 1-57 and over the entire study (days 1-71).
  The highest number of patients among all weeks for the analysis is chosen for each arm.
  Descriptive statistics have been used for this secondary end point.
Time Frame: From baseline to week 10
Measure: Mean (Standard Error); unit: percent days
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 55 | 55
percent days
  Days 1-8 (baseline-week 1) | -138.9 (5.48) | -139.1 (5.67)
  Days 8-15 (week 1-week 2) | -341.9 (9.9) | -328.3 (10.98)
  Days 15-22 (week 2-week 3) | -416.0 (12.06) | -399.8 (14.46)
  Days 22-29 (week 3-week 4) | -447.3 (9.24) | -427.0 (9.76)
  Days 1-29 (baseline-week 4) | -1332.5 (30.78) | -1311.6 (26.35)
  Days 1-57 (baseline-week 8) | -2515.9 (96.98) | -2387.6 (77.61)
  Days 1-71 (baseline-week 10) | -2562.9 (171.86) | -2500.3 (116.10)

6. Secondary Outcome: Еfgartigimod IV and PH20 SC Serum Pharmacokinetic Parameter Ctrough
Description: Evaluation of observed predose concentration (Ctrough) (after all doses for the IV and SC treatment arms). The analysis will present data from Week 1 to Week 4.
  Descriptive statistics have been used for this secondary end point.
Time Frame: From Week 1 to Week 4.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 49 | 51
μg/mL
  Ctrough week 1 | 18.3 (8.05) | 16.4 (33.0)
  Ctrough week 2 | 21.4 (8.36) | 14.0 (6.92)
  Ctrough week 3 | 22.5 (9.61) | 15.2 (8.05)
  Ctrough week 4 | 22.0 (8.12) | 14.9 (6.43)

7. Secondary Outcome: Efgartigimod IV Serum Pharmacokinetic Parameter Cmax
Description: Evaluation of maximum observed concentration (Cmax) (after all doses for the IV treatment arm). The analysis will present data from Baseline to Week 3.
  Descriptive statistics have been used for this secondary end point.
Time Frame: From Baseline to Week 3
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Efgartigimod IV
Number analyzed (Participants) | 54
μg/mL
  Cmax Baseline | 199 (62.8)
  Cmax week 1 | 215 (63.0)
  Cmax week 2 | 211 (75.0)
  Cmax week 3 | 206 (59.5)

8. Secondary Outcome: Incidence of ADA Against Efgartigimod (Safety Analysis Set)
Description: Incidence of antidrug antibodies (ADA) against Efgartigimod in the overall population. ADA analysis is performed with a validated ELISA in a 3-tiered approach (ADA screening analysis, confirmatory analysis and a titration assay). Descriptive statistics have been used for this secondary end point.
Time Frame: From baseline to week 10
Measure: Number; unit: Percent of patients
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 55 | 55
Percent of patients | 34.5 | 20.0

9. Secondary Outcome: Incidence of Antibodies Against rHuPH20 in the SC Treatment Arm (Safety Analysis Set)
Description: Incidence of antibodies against rHuPH20 in the Efgartigimod PH20 SC Arm. antibody analysis is performed with a validated ELISA in a 3-tiered approach (screening analysis, confirmatory analysis and a titration assay) Descriptive statistics have been used for this secondary end point.
Time Frame: From baseline to week 10
Measure: Number; unit: Percent of patients
Arm/Group | Efgartigimod PH20 SC
Number analyzed (Participants) | 55
Percent of patients | 5.5

10. Secondary Outcome: Incidence and Severity of AEs and SAEs (Safety Analysis Set)
Description: Evaluation of incidence and severity of treatment-emergent adverse events (TEAEs) and incidence of serious AEs (SAEs).
  Descriptive statistics have been used for this secondary end point.
Time Frame: From baseline to week 10
Measure: Number; unit: Percent of patients
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 55 | 55
Percent of patients
  ≥1 AE | 67.3 | 50.9
  ≥1 SAE | 14.5 | 7.3
  ≥1 Grade 3 or higher AE | 16.4 | 7.3
  ≥1 AESI | 18.2 | 16.4
  ≥1 Injection site reaction (localized) | 38.2 | 1.8
  ≥1 Infusion- or injection-related reaction | 25.5 | 3.6
  ≥1 Fatal AE | 0 | 0
  ≥1 Treatment-related AE according to PI | 43.6 | 21.8
  ≥1 Procedure-related AE according to PI | 25.5 | 3.6
  ≥1 Treatment-related SAE | 0 | 0
  ≥1 AE for which the IMP was interrupted | 1.8 | 0
  ≥1 AE for which the IMP was discontinued | 3.6 | 0

11. Secondary Outcome: MG-ADL Responders (ITT Analysis Set)
Description: Evaluation of number and percentage of Myasthenia Gravis Activities of Daily Living (MG-ADL) responders in the overall population. The MG-ADL is an 8-item patient-reported scale that assesses MG symptoms and their effects on daily activities. It evaluates a participant's capacity to perform different activities in their daily life, including talking, chewing, swallowing, breathing, brushing their teeth, combing their hair, or getting up from a chair. The MG-ADL also assesses double vision and eyelid droop. It is a discrete quantitative variable in which the 8 items are rated by the participant on a scale of 0 to 3. The total score can range from 0 to 24, with higher total scores indicating more impairment. A participant was considered a MG-ADL responder if he/she showed a reduction of at least 2 points from baseline on the MG-ADL score for at least 4 consecutive weeks. Descriptive statistics have been used for this secondary end point.
Time Frame: From baseline to week 10
Measure: Number; unit: percent
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 55 | 55
percent | 69.1 | 69.1

12. Secondary Outcome: QMG Responders (ITT Analysis Set)
Description: Evaluation of number and percentage of Quantitative Myasthenia Gravis (QMG) responders in the overall population (ITT Analysis Set).
  Descriptive statistics have been used for this secondary end point. One subject in the EFG IV arm had no post-baseline QMG assessment and thus was excluded from the denominator.
Time Frame: From Baseline to Week 10
Population: One patient from Efgartigimod IV didn't have any post-baseline QMG assessment.
Measure: Number; unit: percent
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 55 | 54
percent | 65.5 | 51.9

13. Secondary Outcome: Change From Baseline in MG-ADL Total Score Over Time (ITT Analysis Set)
Description: Evaluation of MG-ADL Total Score Change from baseline over time for the overall population (ITT Analysis Set). Descriptive statistics have been used for this secondary end point.
  The MG-ADL is an 8-item patient-reported scale that assesses MG symptoms and their effects on daily activities. It evaluates a participant's capacity to perform different activities in their daily life, including talking, chewing, swallowing, breathing, brushing their teeth, combing their hair, or getting up from a chair. The MG-ADL also assesses double vision and eyelid droop. It is a discrete quantitative variable in which the 8 items are rated by the participant on a scale of 0 to 3. The total score can range from 0 to 24, with higher total scores indicating more impairment. A participant was considered a MG-ADL responder if he/she showed a reduction of at least 2 points from baseline on the MG-ADL score for at least 4 consecutive weeks.
Time Frame: From baseline to week 10
Measure: Mean (Standard Error); unit: Total score on a scale
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 55 | 55
Total score on a scale
  Week 1 | -2.2 (0.33) | -2.0 (0.30)
  Week 2 | -3.6 (0.40) | -3.2 (0.35)
  Week 3 | -4.7 (0.36) | -4.3 (0.33)
  Week 4 | -5.1 (0.38) | -4.7 (0.37)
  Week 5 | -4.9 (0.36) | -4.3 (0.41)
  Week 6 | -4.2 (0.35) | -3.7 (0.44)
  Week 7 | -3.9 (0.35) | -3.6 (0.44)
  Week 8 | -3.3 (0.34) | -2.9 (0.4)
  Week 10 | -2.2 (0.44) | -2.1 (0.43)

14. Secondary Outcome: Change From Baseline in QMG Score Over Time (ITT Analysis Set)
Description: Evaluation of QMG Total Score change from baseline over time for the overall population (ITT Analysis Set). The QMG (Quantitative Myasthenia Gravis) quantifies disease severity based on impairments of body function and structures as defined by the International Classification of Functioning, Disability and Health. The QMG consists of 13 items that assess ocular, bulbar, and limb function. Six of the 13 items are timed endurance tests measured in seconds. Each item has a possible score from 0 to 3. The total possible score is 39, where higher total scores indicate more severe impairments. It is based on qualitative testing of specific muscle groups to assess limb function.
  Descriptive statistics have been used for this secondary end point. A participant was considered a QMG responder if he/she showed a reduction of at least 3 points from baseline on the QMG score for at least 4 consecutive weeks.
Time Frame: From baseline to week 10
Measure: Mean (Standard Error); unit: Total score
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
Number analyzed (Participants) | 55 | 55
Total score
  Week 1 | -3 (0.48) | -2 (0.44)
  Week 2 | -4.3 (0.58) | -3.4 (0.44)
  Week 3 | -5.7 (0.61) | -4.5 (0.5)
  Week 4 | -6.1 (0.62) | -5.2 (0.52)
  Week 5 | -5.9 (0.61) | -5 (0.57)
  Week 6 | -5.2 (0.6) | -5 (0.61)
  Week 7 | -3.9 (0.61) | -4.1 (0.55)
  Week 8 | -3.7 (0.66) | -3.3 (0.53)
  Week 10 | -2.3 (0.6) | -2.8 (0.53)

ADVERSE EVENTS:
Time Frame: up to 12 weeks (throughout the treatment period)
Description: AEs will be reported by the participant (or, when appropriate, by a caregiver, surrogate, legally authorized representative). The investigator are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study intervention or study procedures, or that caused the participant to discontinue the study intervention.
Groups:
- Efgartigimod IV: Patients receiving efgartigimod intravenous (IV) treatment
  efgartigimod IV: Intravenous infusion of efgartigimod
Arm/Group | Efgartigimod PH20 SC | Efgartigimod IV
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 8/55 | 4/55
Other Adverse Events (participants affected / at risk) | 37/55 | 23/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efgartigimod PH20 SC (N=55) | Efgartigimod IV (N=55)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 5 (5) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Testicular cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efgartigimod PH20 SC (N=55) | Efgartigimod IV (N=55)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 7 (10) | 7 (11)
Myasthenia gravis (Nervous system disorders) | 6 (8) | 1 (2)
Fatigue (General disorders) | 2 (2) | 3 (3)
Injection site bruising (General disorders) | 4 (4) | 0 (0)
Injection site erythema (General disorders) | 7 (7) | 0 (0)
Injection site pain (General disorders) | 3 (3) | 0 (0)
Injection site pruritus (General disorders) | 5 (5) | 0 (0)
Injection site rash (General disorders) | 8 (14) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT04735432/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT04735432/SAP_001.pdf